CLINICAL TRIAL: NCT01812174
Title: On-X Heart Valve - 17mm Aortic and 23mm Mitral
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was terminated due to low/slow enrollment.
Sponsor: On-X Life Technologies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2010-01; G120115 (Other: FDA)
Record Dates: First submitted 2013-03-12; First posted 2013-03-18 (Estimated); Results first posted 2024-03-06 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-02

CONDITIONS: Heart Valve Disease
Keywords: heart valve
MeSH Terms: conditions — Heart Valve Diseases

STUDY DESIGN:
Intervention Model Description: Patients in one arm are recipients of the 17mm On-X Aortic Valve. Patients in the second arm are recipients of the 23mm On-X Mitral Valve. Since double valve cases are exclusionary, these two arms are mutually exclusive and non-randomized.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 17mm On-X Aortic Heart Valve (Experimental): Patients receiving the 17mm On-X aortic heart valve as a replacement for diseased native or prosthetic aortic heart valve.
  Interventions: Device: 17mm aortic valve (On-X )
- 23mm On-X Mitral Heart Valve (Experimental): Patients receiving the 23mm On-X mitral heart valve as a replacement for diseased native or prosthetic mitral heart valve.
  Enrollment into the 23mm On-X mitral arm has been terminated.
  Interventions: Device: 23mm mitral valve (On-X)

INTERVENTIONS:
Device: 17mm aortic valve (On-X ) — Heart aortic valve replacement surgery: 17mm Aortic
  Other Names: On-X prosthetic heart valve
  Arms: 17mm On-X Aortic Heart Valve
Device: 23mm mitral valve (On-X) — Heart mitral valve replacement surgery: 23mm Mitral
  Other Names: On-X prosthetic heart valve
  Arms: 23mm On-X Mitral Heart Valve

SUMMARY:
This study examines the hemodynamic and hemolytic properties of two additional smaller size valves to the On-X line of valves already approved by FDA.

DETAILED DESCRIPTION:
The purpose of the study is to assess the safety and efficacy of the 17mm On-X Aortic Prosthetic Heart Valve and the 23mm On-X Mitral Prosthetic Heart Valve when used to replace diseased aortic or mitral valves in human subjects.

The On-X 17mm aortic valve will be implanted in approximately 20 and at least 15 patients who will be followed for at least 1 year. Patients will be any age and will require this size valve as determined in surgery but will be recruited prior to surgery based on results of preoperative screening tests.

Enrollment into the 23mm mitral arm of the study has been terminated.

ELIGIBILITY:
Inclusion Criteria:

1. Patients of any age; unless waived by local IRB assent of the patient and in all cases consent of parent or legally authorized representative is required if a patient is under the age of majority and not legally emancipated.
2. Patients who are sufficiently ill to warrant replacement of their diseased natural or prosthetic valve, based on standard cardiovascular diagnostic workups.
3. Patients who are in sufficient satisfactory condition, based on the physical exam and investigator's experience, to be an average or better operative risk, (i.e., likely to survive one year postoperatively).
4. Patients who require an isolated aortic valve replacement size 17 mm or isolated mitral valve replacement size 23mm.
5. Patients who are geographically stable and willing to return to the implanting center for follow-up visits.
6. Patients or legally authorized representatives who are adequately informed of their participation in the clinical study and what will be required of them in order to comply with the protocol.
7. Patients requiring concomitant cardiovascular surgery, such as coronary bypass may be included in the study.

Exclusion Criteria:

1. Patients who are pregnant, planning to become pregnant or are lactating. 2 Patients who have a noncardiac progressive disease, which in the investigator's experience produces an unacceptable increased risk to the patient.

3 Patients who have a documented history of substance (drug or alcohol) abuse or are prison inmates.

4. Patients with a previous prosthetic valve, where it is not being replaced by a study valve, or patients requiring multiple valve replacement.

5. Patients with active endocarditis or active myocarditis. 6 Patients who require tricuspid or pulmonic valve replacement. 7. Patients who have not agreed to return for the required number of follow-up visits or who are geographically unavailable for follow-up.

8. Patients who cannot be maintained on long-term anticoagulant therapy. 9. Patients with non-cardiac illness resulting in a life expectancy of less than 1-year.

10. Patients previously enrolled and implanted in this trial may not re-enter after withdrawal.

11. Patients already enrolled in another investigational device or drug study (nor can enrolled patients be enrolled in other studies).

12. Patients with acute preoperative neurological deficit, myocardial infarction, or cardiac event who have not returned to baseline for at least 30-days prior to enrollment.

13. Patients with aortic aneurysm or other medical condition that creates a higher than usual risk of surgical complication.

14. Patients who are prisoners or mentally ill, and pediatric patients who are incapable of understanding their assent as judged by the principal investigator.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-11-18 (Actual); Primary Completion 2018-12-07 (Actual); Study Completion 2018-12-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sidney Levitsky, MD, Study Chair — Beth Israel Deaconess Medical Center
Locations (10):
- United States (7):
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Maine Medical Center, Portland, Maine
  - Children's Heart Center Nevada, Las Vegas, Nevada
  - Cincinnati Children's Medical Center, Cincinnati, Ohio
  - University of Oklahoma/Children's Hospital, Oklahoma City, Oklahoma
  - University of Virginia, Charlottesville, Virginia
  - Mary Bridge Children's - Tacoma General Hospital, Tacoma, Washington
- Mayaguez Medical Center, Mayagüez, PR, Puerto Rico
- Spain (2):
  - Hospital Clinico Provincial, Barcelona
  - University Hospital Salamanca, Salamanca

RESULTS

PARTICIPANT FLOW:
Groups:
- 23mm On-X Mitral Heart Valve: Patients receiving the 23mm On-X mitral heart valve as a replacement for diseased native or prosthetic mitral heart valve.
  23mm mitral valve (On-X): Heart mitral valve replacement surgery: 23mm Mitral
Period: Overall Study
Arm/Group | 17mm On-X Aortic Heart Valve | 23mm On-X Mitral Heart Valve
Started | 14 | 6
Completed | 11 | 6 (The 23mm Mitral Arm of the study was terminated early, see approval letter G120115/S005 dated Nov 16, 2017. All subjects in this arm were followed until completion of their normal follow-up schedule.)
Not Completed | 3 | 0
Not completed — Death | 1 | 0
Not completed — Protocol Violation | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 17mm On-X Aortic Heart Valve | 23mm On-X Mitral Heart Valve | Total
Number analyzed (Participants) | 14 | 6 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2 | 5 | 7
  Between 18 and 65 years | 2 | 1 | 3
  >=65 years | 10 | 0 | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 3 | 14
  Male | 3 | 3 | 6
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Puerto Rico | 5 | 0 | 5
  United States | 4 | 6 | 10
  Spain | 5 | 0 | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Valve Related Adverse Events at 1 Year
Description: Number of subjects with a valve related adverse event at 1 year.
Time Frame: 1 Year
Population: All adverse events for all enrolled subjects, regardless of study completion are counted.
Measure: Count of Participants; unit: Participants
Arm/Group | 17mm On-X Aortic Heart Valve | 23mm On-X Mitral Heart Valve
Number analyzed (Participants) | 14 | 6
Participants | 0 | 0

2. Secondary Outcome: Diagnosis of Valve Thrombosis at 1 Year
Description: Number of subjects with a diagnosis of Valve Thrombosis at 1 year
Time Frame: 1-year
Population: Only subjects that completed the 1 year follow up were included in this analysis.
Measure: Count of Participants; unit: Participants
Groups:
- 23mm On-X Mitral Heart Valve: Patients receiving the 23mm On-X mitral heart valve as a replacement for diseased native or prosthetic mitral heart valve.
  Enrollment into the 23mm On-X mitral arm has been terminated.
  23mm mitral valve (On-X): Heart mitral valve replacement surgery: 23mm Mitral
Arm/Group | 17mm On-X Aortic Heart Valve | 23mm On-X Mitral Heart Valve
Number analyzed (Participants) | 11 | 6
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from time of implant up to 1 year post implant.
Arm/Group | 17mm On-X Aortic Heart Valve | 23mm On-X Mitral Heart Valve
All-Cause Mortality (participants affected / at risk) | 2/14 | 0/6
Serious Adverse Events (participants affected / at risk) | 6/14 | 1/6
Other Adverse Events (participants affected / at risk) | 0/14 | 0/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 17mm On-X Aortic Heart Valve (N=14) | 23mm On-X Mitral Heart Valve (N=6)
Permanent Pacemaker Implant (Cardiac disorders) | 2 (2) | 1 (1)
Dislocation of Right Temporomandibular joint (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
COPD (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Bleed- Major (Surgical and medical procedures) | 2 (4) | 0 (0)
Septic Shock (Infections and infestations) | 1 (1) | 0 (0)
Congestive Heart Failure (Cardiac disorders) | 1 (1) | 0 (0)
Pulmonary Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All information which I hereafter obtain from ON-X LIFE TECHNOLOGIES … about or relating to the prosthesis … which is the subject of this study and all information which I have … concerning this study is considered by ON-X to be proprietary and confidential to ON-X .I … will not use such confidential information, or release, reveal or disclose such confidential information to anyone without the written consent of ON-X or prior public disclosure by ON-X.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-09-29): https://cdn.clinicaltrials.gov/large-docs/74/NCT01812174/Prot_SAP_000.pdf